CLINICAL TRIAL: NCT06261619
Title: A Comparative Trial Between Sotair® Device Attached to Manual Resuscitator Versus Manual Ventilation Alone in Patients Undergoing Non-emergent Surgery With General Anesthesia: A Prospective Randomized Cross-over Clinical Trial
Brief Title: Superiority Trial Between Sotair® Device Attached to Manual Resuscitator Versus Ventilation Alone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Mark Kendall, Director of Clinical Research, Rhode Island Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2079951
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Airway Management; Respiration, Artificial
Keywords: Mechanical Ventilation; General Anesthesia; Bag Mask Ventilation; Adult Sotair Device
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Study Design: A superiority trial; a single two-group cross over randomized trial.
Who Masked: Participant
Masking Description: The care provider will not know the recorded lung function recordings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Bag mask ventilation with Adult Sotair device (Active Comparator): The anesthesia provider will manually bag ventilate with the Adult Sotair® device for 3 minutes with an average respiratory rate of 12 breaths per minute with a deep breath every 30 seconds.
  Interventions: Device: Adult Sotair Device
- Bag mask ventilation (No Intervention): The anesthesia provider will manually bag ventilate for 3 minutes with an average respiratory rate of 12 breaths per minute with a deep breath every 30 seconds.

INTERVENTIONS:
Device: Adult Sotair Device — Adult Sotair® device employs a flow limiting valve mechanism.
  Other Names: Sotair; SafeBVM
  Arms: Bag mask ventilation with Adult Sotair device

SUMMARY:
Effective respiratory ventilation is achieved by moving the right amount of air to and out of the lungs while keeping the pressures at a safe level. A disposable safety device, Adult Sotair®, was created to improve manual ventilation delivery. In this superiority study, the investigators will perform two-group cross over randomized design to test the superiority of the Adult Sotair® device compared to manual ventilation alone.

DETAILED DESCRIPTION:
Poor manual ventilation technique is a well-documented problem which occurs irrespective of a provider's qualifications or experience. A disposable safety device, Adult Sotair®, was created to improve manual ventilation delivery among providers. The device is attached to a bag valve mask (i.e. manual resuscitator) and employs a flow limiting valve mechanism to minimize excessive pressure in the airway system without venting air by capping peak flow rates at 55 L/min. For an average adult with normal lung compliance and resistance, this corresponds to a maximum airway pressure of approximately 20 cmH2O which minimizes air entry into the stomach. In this superiority study, the investigators will use a two-group cross over randomized design to test the superiority of the Adult Sotair® device compared to manual ventilation alone with respect to airway pressure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who are scheduled for non-emergency surgery with general anesthesia (w/artificial airway) at Rhode Island Hospital.
* American Society Of Anesthesiologists Physical Status 1 and 2

Exclusion Criteria:

* American Society of Anesthesiologists Physical Status >3 (e.g. respiratory disease)
* Oropharyngeal or facial pathology

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
Peak airway pressure | Recorded every thirty seconds for a total duration of 3 minutes for each arm of the study
  Mean of the maximum peak airway pressures expressed in cm H2O

SECONDARY OUTCOMES:
Tidal volume | Recorded every thirty seconds for a total duration of 3 minutes for each arm of the study
  The amount of air that moves to or out of the lungs with each respiratory cycle. Measured in mL. Mean of the maximum tidal volumes every 30 seconds.
Airflow | Recorded every thirty seconds for a total duration of 3 minutes for each arm of the study
  Represents the volume of air moved per unit of time during inspiration and expiration. Measured (L/min)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kendall, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
The IPD that underlie the results in a publication will be shared with other researchers.
Supporting Information: SAP
Time Frame: The SAP will be available at the end of the trial for three years. The data that supports the findings of the study will be available form the corresponding investigator upon reasonable request.

REFERENCES:
- [Background] Fogarty M, Kuck K, Orr J, Sakata D. A comparison of controlled ventilation with a noninvasive ventilator versus traditional mask ventilation. J Clin Monit Comput. 2020 Aug;34(4):771-777. doi: 10.1007/s10877-019-00365-1. Epub 2019 Jul 23. PMID 31338661
- [Background] von Goedecke A, Bowden K, Wenzel V, Keller C, Gabrielli A. Effects of decreasing inspiratory times during simulated bag-valve-mask ventilation. Resuscitation. 2005 Mar;64(3):321-5. doi: 10.1016/j.resuscitation.2004.09.003. PMID 15733761
- [Background] Culbreth RE, Gardenhire DS. Manual bag valve mask ventilation performance among respiratory therapists. Heart Lung. 2021 May-Jun;50(3):471-475. doi: 10.1016/j.hrtlng.2020.10.012. Epub 2020 Nov 1. PMID 33138977
- See also: Adult Sotair Products — https://safebvm.com/